CLINICAL TRIAL: NCT01315548
Title: Contrast Enhanced Harmonic Endoscopic Ultrasound (CEH-EUS) Used in the Differentiation of Focal Pancreatic Masses
Brief Title: Contrast Enhanced Harmonic Endoscopic Ultrasound (CEH-EUS) in Focal Pancreatic Masses
Status: Completed | Type: Observational
Sponsor: University of Medicine and Pharmacy Craiova (Other)
Collaborators: Copenhagen University Hospital, Denmark (Other); Caritas-Krankenhaus Bad Mergentheim (Other); Institut Paoli-Calmettes (Other); University of Witten/Herdecke (Other); Hospital Meiningen Germany (Unknown); Odense University Hospital (Other); University of Santiago de Compostela (Other); Università Vita-Salute San Raffaele (Other); SRH Wald-Klinikum Gera GmbH (Other); University of Bergen (Other); Institutul Clinic Fundeni (Other); Glasgow Royal Infirmary (Other); University College, London (Other)
Responsible Party: Sponsor
Other Study IDs: CEH-EUS-001; CEH-EUS-UMFCV-RO
Record Dates: First submitted 2011-03-13; First posted 2011-03-15 (Estimated); Last update posted 2018-01-17 (Actual); Status verified 2018-01

CONDITIONS: Adenocarcinoma Pancreas; Chronic Pancreatitis
Keywords: Contrast enhanced harmonic endoscopic ultrasound; Pancreatic adenocarcinoma; Chronic pancreatitis
MeSH Terms: conditions — Pancreatitis, Chronic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Pathology samples obtained from duodeno-pancreatectomies or caudal pancreatectomies done with curative intent, as well as microhistological fragments obtained through EUS-FNA biopsy processed by paraffin embedding
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Pancreatic adenocarcinoma: Patients diagnosed with solid pancreatic adenocarcinoma masses, with cytological / histologicalconfirmation
- Chronic pancreatitis: Patients diagnosed with solid pancreatic tumor masses with all the criteria fulfilled to exclude pancreatic cancer

SUMMARY:
The aim of the study is to assess the accuracy of real-time perfusion imaging pattern of pancreatic focal lesions visualized by contrast-enhanced harmonic endoscopic ultrasound (CEH-EUS) for the differential diagnosis between chronic pseudotumoral pancreatitis and pancreatic cancer in a prospective multicenter design.

The study will include patients with focal pancreatic masses evaluated by CEH-EUS and EUS-FNA. The diagnosis is usually unknown in the moment of the initial evaluation, the patients being included based on a suspicion of focal pancreatic masses after transabdominal ultrasound, CT or MR examinations. However, after a complete evaluation, a final diagnosis will be reached based on the combination of EUS-FNA cytology/pathology, surgical pathology and minimum 12 months follow-up.

DETAILED DESCRIPTION:
Ultrasound contrast agents in conjunction with contrast specific imaging techniques are increasingly accepted in clinical use for diagnostic imaging. The study of the pancreas is a new and promising application of contrast-enhanced ultrasound (CE-US), including contrast-enhanced endoscopic ultrasound (CE-EUS). The technique is not indicated to improve the detection of pancreatic lesions, but to improve the delineation and differential diagnosis of pancreatic lesions. One of the fluoro-gas-containing contrast agents used in CE-US and CE-EUS is Sonovue®, which consists of phospholipids-stabilized bubbles of sulfurhexafluoride (SF6). Sonovue® is isotonic, stable and resistant to pressure, with a viscosity similar to blood. It does not diffuse into the extravascular compartment remaining within the blood vessels until the gas dissolves and is eliminated in the expired air (blood pool contrast agent). The safety profile of SonoVue showed a very low incidence of side effects; it is not nephrotoxic and the incidence of severe hypersensitivity is similar to other magnetic resonance imaging contrast agents. Moreover, Sono-Vue is approved for clinical use in EU countries. The blood supply of the pancreas is entirely arterial, making contrast-enhanced examinations feasible and readily available. Based on the European Federation Societies of Ultrasound in Medicine and Biology guidelines and recommendations, updated in 2008, two phases were defined for CE-US and CE-EUS of the pancreas: an early/arterial phase (starting from 10 to 30 seconds) and a venous/late phase (from 30 to 120 seconds).

Distinguishing pancreatic adenocarcinoma from other pancreatic masses remains challenging with current imaging techniques. The specificity of the discrimination between benign and malignant focal pancreatic lesions was found to be 93.3% using power Doppler contrast-enhanced EUS (PD-CE-EUS) compared with 83.3% for conventional EUS. The hypovascular aspect of lesions under PD-CE-EUS seemed highly sensitive and specific (higher than 90%) for adenocarcinoma in several published studies. During PD-CE-EUS examinations the ultrasound frequency returned to the transducer is the same with that transmitted, but the method is associated with artifacts resulting from turbulent flow (flash and overpainting). At CE-EUS, ductal adenocarcinoma is typically hypoenhanced compared to the adjacent pancreatic tissue in all phases. Furthermore, the lesion size and margins are better visualized, as well as the relationship with peripancreatic arteries and veins. Focal lesions in chronic pancreatitis are reported to have similar or hyper enhancement features as compared to the normal pancreatic parenchyma.

Dedicated contrast-enhanced harmonic EUS techniques (based on a low mechanical index) are recently available in new EUS systems. The harmonic frequencies returned during CEH-EUS are different from those transmitted by the transducer and are the result of non-linear oscillations of the microbubbles. The image obtained is an addition of the signal created by the distortion of the microbubbles and the tissue-derived signal. This can be optimized by using low MI, which allows minimum bubble destruction and complete "subtraction" of the tissue derived signal, obtaining a high resolution continuous real-time assessment of the microvascularization during the contrast uptake period (real-time perfusion imaging). CEH-EUS allows a more precise location of vascular structures within the parenchyma and focal abnormalities, with better delineation of pancreatic lesions than EUS, especially in the cases where air or fat causes artifacts and insufficient visualization of the pancreatic parenchyma. An initial pilot study described an experimental technique of CEH-EUS based on a linear prototype EUS scope, a low mechanical index (0.08 - 0.25) and a 2nd generation contrast agent (Sono-Vue), which allowed the visualization of early arterial phase and late parenchymal phase enhancement of the pancreas. Another pilot study demonstrated both real-time continuous images of finely branching vessels of the pancreas and intermittent homogenous parenchymal perfusion images, by using a radial prototype EUS scope, a low mechanical index (0.4) and a 2nd generation contrast agent (Sono-Vue). Several other research groups already reported the feasibility of CEH-EUS with low mechanical index. The sensitivity, specificity and accuracy for diagnosing pancreatic adenocarcinoma were 88%, 89%, and 88.5% in one study and 80%, 91.7%, and 86% in the other study. However, the data is still limited and a prospective, multicentric blinded study would certainly be necessary.

The study design is prospective, blinded and multi-center, comparing contrast-enhanced harmonic endoscopic ultrasound (CEH-EUS) results for the detection and characterization of focal pancreatic masses, in comparison with the gold standard represented by pathology. The study will be performed with the approval of the institutional board review of each center. The study protocol will be uploaded on ClinicalTrials.gov, the registry of federally and privately supported clinical trials conducted in the United States and around the world.

The study is already approved by the ethical committee of the University of Medicine and Pharmacy Craiova, Romania (attached). According to EFSUMB (European Federation Societies for Ultrasound in Medicine and Biology) guidelines published in 2008, second-generation contrast agents are also approved in the E.U. for ultrasound examinations, including liver and pancreas examinations.

All patients with a suspicion (clinical, US, CT/MR) of pancreatic masses should undergo EUS, contrast-enhanced harmonic EUS and EUS-elastography, as well as EUS-FNA

EUS with EUS-guided FNA

* Protocol of EUS with EUS-FNA should include linear EUS instruments with complete examinations of the pancreas.
* Tumor characteristics (echogenicity, echostructure, size) will be described as well as presence / absence of power Doppler signals.
* EUS-FNA will be performed in all pancreatic masses with at least three passes
* All examiners should be blinded for the results of pathology

CEH-EUS procedure

* A two panel image with the usual conventional gray-scale B-mode EUS image on the right side and with the contrast harmonic image on the left side will be used, according to pre-established presets.
* A low mechanical index procedure (dynamic wide-band contrast harmonic imaging mode) will be used, with a mechanical index of 0.08-0.25 and corresponding powers.
* The starting point of the timer will be considered the moment of intravenous contrast injection (Sonovue 4.8 mL).
* CEH-EUS will be performed during usual EUS examinations, with the whole movie (T0-T120s) recorded on the embedded HDD of the ultrasound system, for later analysis.
* In order to minimize human bias, all post-processing and computer analysis of digital movies will be performed within the coordinating IT Center, with all programmers and statisticians being blinded to the clinical, imaging and pathological data.

EUS-elastography procedures

* An additional EUS elastography movie of 30 seconds should be saved on the embedded HDD.
* The following settings will be used for EUS elastography: examination frequency is usually set at 7.5 MHz, while preinstalled system settings are used in all patients: reject (2), E-smoothing (2), persistence (3), and E-dynamic range (4).

Final diagnosis The diagnosis of chronic pancreatitis will be based on the clinical information (history of alcohol abuse, previous diagnosis of chronic pancreatitis or diabetes mellitus), as well as a combination of imaging methods (ultrasound, CT and EUS). At least four criteria of chronic pancreatitis during EUS will be considered for the positive diagnosis. The diagnosis of chronic pseudotumoral pancreatitis will always be confirmed by surgery or by a follow-up of at least six months used to exclude malignancy in the patients that will not be operated on.

A positive cytological diagnosis will be taken as a final proof of malignancy of the pancreas mass. The diagnoses obtained by EUS-FNA will be further verified either by surgery or during a clinical follow-up of at least 6 months.

Pathology samples obtained from duodeno-pancreatectomies or caudal pancreatectomies done with curative intent, as well as microhistological fragments obtained through EUS-FNA biopsy will be processed by paraffin embedding with usual colorations (haematoxylin-eosin), with subsequent immune-histochemistry at the discretion of the participating centers pathologists in order to exclude neuroendocrine tumors / pancreatic metastases.

The patients will be followed-up for at least six months through clinical examination, biological exams and transabdominal ultrasound, eventually with a repeat spiral CT / EUS after six months.

Statistical analysis All results will be expressed as mean ± standard deviation (SD). Differences between the patients with pancreatic cancer and chronic pancreatitis will performed by the two-sample t-test (two independent samples). Since this parametric method makes assumptions about normality and similar variances, we will initially perform both the Kolmogorov-Smirnov and Shapiro-Wilk W normality tests and verify the equality of variances assumption with the F test. In the case of the two-sample t-test, we will also perform the non-parametric alternative given by the Mann-Whitney U test, since in some instances it may even offer greater power to reject the null hypothesis than the t-test.

Since with more than two groups of observations it is far better to use a single analysis that enables us to look at all the data in the same time, we will also perform the one-way analysis of variance (ANOVA) method with the same baseline assumptions. A p-value less than 0.05 will be considered as statistically significant.

Sensitivity, specificity, positive predictive value, negative predictive value and accuracy of CEH-EUS +/- will be determined in comparison with the final diagnosis.

The estimated number of patients included is at least 210, based on at least 10 centers with at least 20 patients each, which will be enrolled in an 18 months period. The power analysis was based on the following assumption: in order to use the powerful t-test for independent samples, a sample size equaling 105 patients in each group is sufficient to provide 95% statistical power to detect a difference of 5% in mean, for a type I error alpha = 0.05, and the population standard deviation = 10%. The difference in mean was based on previously published data which report an accuracy of approximately 80-85% for EUS-FNA, and 90% for contrast-enhanced EUS.

ELIGIBILITY:
Inclusion Criteria:

* Patients with suspicion of solid pancreatic tumor masses by previous cross-sectional imaging techniques (US, CT, MR)
* Age 18 to 90 years old, men or women
* Signed informed consent for EUS with contrast-enhancement, elastography and EUS-FNA

Exclusion Criteria:

* Prior surgical treatment with curative intent or chemo-radiotherapy
* Patients diagnosed with mucin producing tumors, pancreatic cystic tumors, etc.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The diagnosis of chronic pancreatitis will be based on the clinical information (history of alcohol abuse, previous diagnosis of chronic pancreatitis or diabetes mellitus), as well as a combination of imaging methods (ultrasound, CT and EUS). At least four criteria of chronic pancreatitis during EUS will be considered for the positive diagnosis.
  A positive cytological diagnosis will be taken as a final proof of malignancy of the pancreas mass. The diagnoses obtained by EUS-FNA will be further verified either by surgery or during a clinical follow-up of at least 6 months.
Sampling Method: Non-Probability Sample
Enrollment: 210 (Actual)
Dates: Start 2011-03; Primary Completion 2012-04 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Contrast enhanced harmonic endoscopic ultrasound | Every six months
  Value of contrast enhanced harmonic endoscopic ultrasound for the differential diagnoses of pancreatic masses.

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Săftoiu, Professor, Study Director — University of Medicine and Pharmacy Craiova, Romania
Locations (14):
- Denmark (2):
  - Department of Surgical Gastroenterology, Gentofte & Herlev Hospital, University of Copenhagen, Copenhagen
  - Center for Surgical Ultrasound, Department of Surgery, Odense University Hospital, Odense
- Paoli-Calmettes Institut, Marseille, France
- Germany (4):
  - Caritas-Krankenhaus Bad Mergentheim, Bad Mergentheim
  - SRH Wald-Klinikum, Gera
  - Department of Internal Medicine II, Hospital Meiningen, Meiningen
  - Helios Klinikum, University of Witten/Herdecke, Wuppertal
- Gastroenterology and Gastrointestinal Endoscopy Unit, Vita Salute San Raffaele University, Milan, Italy
- Insitute of Medicine, University of Bergen and National Centre for Ultrasound in Gastroenterology, Haukeland University Hospital, Bergen, Norway
- Romania (2):
  - Center of Gastroenterology and Hepatology, Fundeni Clinical Institute, Bucharest
  - Gastroenterology Department, University of Medicine and Pharmacy, Craiova
- University Hospital, Santiago de Compostela, Santiago de Compostela, Spain
- United Kingdom (2):
  - Hepatobiliary Surgery, Glasgow Royal Infirmary, Glasgow
  - Institute of Hepatology, University College London, London

REFERENCES:
- [Background] Claudon M, Cosgrove D, Albrecht T, Bolondi L, Bosio M, Calliada F, Correas JM, Darge K, Dietrich C, D'Onofrio M, Evans DH, Filice C, Greiner L, Jager K, Jong Nd, Leen E, Lencioni R, Lindsell D, Martegani A, Meairs S, Nolsoe C, Piscaglia F, Ricci P, Seidel G, Skjoldbye B, Solbiati L, Thorelius L, Tranquart F, Weskott HP, Whittingham T. Guidelines and good clinical practice recommendations for contrast enhanced ultrasound (CEUS) - update 2008. Ultraschall Med. 2008 Feb;29(1):28-44. doi: 10.1055/s-2007-963785. No abstract available. PMID 18270887
- [Background] Seicean A, Badea R, Stan-Iuga R, Gulei I, Pop T, Pascu O. The added value of real-time harmonics contrast-enhanced endoscopic ultrasonography for the characterisation of pancreatic diseases in routine practice. J Gastrointestin Liver Dis. 2010 Mar;19(1):99-104. PMID 20361085
- [Background] Hocke M, Schulze E, Gottschalk P, Topalidis T, Dietrich CF. Contrast-enhanced endoscopic ultrasound in discrimination between focal pancreatitis and pancreatic cancer. World J Gastroenterol. 2006 Jan 14;12(2):246-50. doi: 10.3748/wjg.v12.i2.246. PMID 16482625
- [Background] Saftoiu A, Iordache SA, Gheonea DI, Popescu C, Malos A, Gorunescu F, Ciurea T, Iordache A, Popescu GL, Manea CT. Combined contrast-enhanced power Doppler and real-time sonoelastography performed during EUS, used in the differential diagnosis of focal pancreatic masses (with videos). Gastrointest Endosc. 2010 Oct;72(4):739-47. doi: 10.1016/j.gie.2010.02.056. Epub 2010 Aug 2. PMID 20674916
- [Background] Seicean A. Endoscopic ultrasound in chronic pancreatitis: where are we now? World J Gastroenterol. 2010 Sep 14;16(34):4253-63. doi: 10.3748/wjg.v16.i34.4253. PMID 20818808
- [Background] Dietrich CF, Ignee A, Frey H. Contrast-enhanced endoscopic ultrasound with low mechanical index: a new technique. Z Gastroenterol. 2005 Nov;43(11):1219-23. doi: 10.1055/s-2005-858662. PMID 16267707
- [Background] Seicean A, Badea R, Stan-Iuga R, Mocan T, Gulei I, Pascu O. Quantitative contrast-enhanced harmonic endoscopic ultrasonography for the discrimination of solid pancreatic masses. Ultraschall Med. 2010 Dec;31(6):571-6. doi: 10.1055/s-0029-1245833. Epub 2010 Nov 15. PMID 21080306
- [Derived] Saftoiu A, Vilmann P, Dietrich CF, Iglesias-Garcia J, Hocke M, Seicean A, Ignee A, Hassan H, Streba CT, Ioncica AM, Gheonea DI, Ciurea T. Quantitative contrast-enhanced harmonic EUS in differential diagnosis of focal pancreatic masses (with videos). Gastrointest Endosc. 2015 Jul;82(1):59-69. doi: 10.1016/j.gie.2014.11.040. Epub 2015 Mar 16. PMID 25792386
- See also: Related Info — http://study.umfcv.ro/ceh-eus-pancreas/